CLINICAL TRIAL: NCT00266071
Title: Study of the Cutaneous Microcirculation in Elderly People
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Other Study IDs: PHRC05-08
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-12

CONDITIONS: Elderly People
Keywords: skin; pressure; age

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Cutaneous response

SUMMARY:
Pressure ulcers are a common and frustrating problem and their treatment is critical in elderly people. The interaction between external pressure and the skin vascular is central to the prevention of pressure ulcers. It is only through understanding of the physiology of cutaneous perfusion and its relation to external pressure or different stimuli that effective preventive measures to reduce skin beakdown can be adapted in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* volunteers

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis SAUMET, MD PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Laboratoire de Physiologie - CHU, Angers, France